CLINICAL TRIAL: NCT02892630
Title: Immune Thrombocytopenia in Pregnancy: Evolution and Prognostic Factors According to a Prospective Observational Comparative Multicenter National French Study
Brief Title: Immune Thrombocytopenia in Pregnancy
Acronym: TIGRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM12204
Record Dates: First submitted 2016-07-31; First posted 2016-09-08 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Immune Thrombocytopenia; Pregnancy
Keywords: Immune Thrombocytopenia; Pregnancy
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pregnant ITP women: Pregnant women more than 18 years old, with primary ITP diagnosis before pregnancy
  Interventions: Other: No intervention
- Control ITP Women (Non pregnant): Primary ITP women more than 18 years old, at more than one year from a precedent pregnancy
  Interventions: Other: No intervention
- De novo ITP pregnant women: Pregnant women more than 18 years old, with newly diagnosed thrombocytopenia during pregnancy
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The pregnancy may activate flares of certain autoimmune diseases such as lupus. The influence of pregnancy on the evolution of ITP was never studied while this pathology affects firstly women old enough to procreate. Also, the influence of ITP on pregnancy (risk of obstetric complications) and on newborns (risk of neonatal thrombocytopenia) is rather unknown and never studied in a prospective study. The realization of a prospective study to answer these questions is necessary to allow us to inform better the patients affected by ITP and to define better in this context the strategy of supervision of the mother, the foetus and the newborn. The highlighting of risk factors of ITP flare or obstetric or neonatal complications will indeed allow the implementation of prevention measures.

The conclusions of this study will allow us to adapt national guidelines for ITP during pregnancy.

ELIGIBILITY:
1. Pregnant ITP women Inclusion Criteria

   * Women more than 18 years old
   * Primary ITP diagnosis, defined according to international criteria of 2009 consensus conference (isolated thrombocytopenia <100 G/L)
   * And pregnancy diagnosis after ITP diagnosis
   * Information notice delivered to women with non opposition to participation to the study Exclusion Criteria
   * Secondary ITP (according to 2009 consensus conference)
   * Severe comorbidity making difficult women's following
2. Control ITP Women (Non pregnant) Inclusion Criteria

   * Women more than 18 years old
   * Primary ITP diagnosis, defined according to international criteria of 2009 consensus conference (isolated thrombocytopenia <100 G/L)
   * Non pregnant (> 12 months of precedent pregnancy)
   * (Matched on age+/- 5 years old: suppress by amendment n°3 20170117), phase and status of ITP, and history of splenectomy
   * Information notice delivered to women with non opposition to participation to the study Exclusion Criteria
   * Secondary ITP (according to 2009 consensus conference)
   * Severe comorbidity making difficult women's following
3. De novo ITP pregnant women Inclusion Criteria

   * Women more than 18 years old
   * Pregnant
   * With a newly diagnosed thrombocytopenia <50G/L, after elimination of others thrombocytopenia etiologies during pregnancy: gestational thrombocytopenia, preeclampsia, HELLP syndrome, ….
   * Information notice delivered to women with non opposition to participation to the study Exclusion Criteria
   * Secondary ITP (according to 2009 consensus conference)
   * Severe comorbidity making difficult women's following
   * Non confirmation of ITP diagnosis in post-partum

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from French referral centers for immune Thrombocytopenia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-02-03 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Composite criteria including in the two principal groups (pregnant and none pregnant) : Frequency of: - ITP treatment modification,- biologic worsening and severe thrombocytopenia (<30G/L), - hemorrhagic complication and ITP status modification | During 15 months (9 months of pregnancy and 6 months of post partum)
  The biologic worsening is defined by a platelet decrease > 30% compared to platelet count before pregnancy

SECONDARY OUTCOMES:
Identification of risk factors of ITP worsening during pregnancy | During 15 months
Evaluation of obstetrical complications in case of ITP | During 15 months
Evaluation of neonatal thrombocytopenia in case of maternal ITP | During 15 months
Identification of the risk factors of obstetrical complications | During 15 months
Identification of the risk factors of neonatal thrombocytopenia | During 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Godeau, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182
- [Background] Fujimura K, Harada Y, Fujimoto T, Kuramoto A, Ikeda Y, Akatsuka J, Dan K, Omine M, Mizoguchi H. Nationwide study of idiopathic thrombocytopenic purpura in pregnant women and the clinical influence on neonates. Int J Hematol. 2002 May;75(4):426-33. doi: 10.1007/BF02982137. PMID 12041677
- [Background] Webert KE, Mittal R, Sigouin C, Heddle NM, Kelton JG. A retrospective 11-year analysis of obstetric patients with idiopathic thrombocytopenic purpura. Blood. 2003 Dec 15;102(13):4306-11. doi: 10.1182/blood-2002-10-3317. Epub 2003 Aug 28. PMID 12947011
- [Background] Valat AS, Caulier MT, Devos P, Rugeri L, Wibaut B, Vaast P, Puech F, Bauters F, Jude B. Relationships between severe neonatal thrombocytopenia and maternal characteristics in pregnancies associated with autoimmune thrombocytopenia. Br J Haematol. 1998 Nov;103(2):397-401. doi: 10.1046/j.1365-2141.1998.01006.x. PMID 9827911
- [Background] Provan D, Stasi R, Newland AC, Blanchette VS, Bolton-Maggs P, Bussel JB, Chong BH, Cines DB, Gernsheimer TB, Godeau B, Grainger J, Greer I, Hunt BJ, Imbach PA, Lyons G, McMillan R, Rodeghiero F, Sanz MA, Tarantino M, Watson S, Young J, Kuter DJ. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood. 2010 Jan 14;115(2):168-86. doi: 10.1182/blood-2009-06-225565. Epub 2009 Oct 21. PMID 19846889